CLINICAL TRIAL: NCT06817395
Title: Prevalence, Reproducibility, and Feasibility of Longitudinal Assessment of Neurocognitive Dysfunction in Adults with Chronic and Persistent Immune Thrombocytopenia (COGFIT)
Brief Title: Cognitive Dysfunction in Chronic and Persistent Immune Thrombocytopenia
Acronym: COGFIT
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Platelet Disorder Support Association (PDSA) (Unknown)
Responsible Party: Principal Investigator, Debbie Jiang, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2024P000181
Record Dates: First submitted 2025-01-28; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Immune Thrombocytopenia
Keywords: Cognitive impairment; Immune thrombocytopenia; ITP; Quality of life; Cognitive dysfunction; Cognition
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults with chronic or persistent ITP

SUMMARY:
Individuals with immune thrombocytopenia (ITP) frequently report difficulties with attention and memory. The main question this study seeks to answer is:

Do patients with ITP have evidence of cognitive impairment as detected by a cognitive function test battery?

To address this issue, participants will take a cognitive function test and complete surveys on quality of life, fatigue, depression, and cognitive symptoms. The primary aim of the study is to evaluate for the presence and extent of cognitive impairment in patients with ITP. The study will also assess whether cognitive impairment in ITP is associated with patient-reported impacts on quality of life, fatigue, mood, and cognitive symptoms as well as clinical characteristics such as ITP disease and treatment history.

DETAILED DESCRIPTION:
This is a longitudinal observational study that seeks to evaluate for the prevalence and extent of cognitive dysfunction in adults with persistent and chronic ITP. Following enrollment, subjects will complete neurocognitive testing using the NIH Toolbox Cognition Battery (NIHTB-CB). In addition, subjects will complete surveys for patient-reported outcomes of quality of life, fatigue, self-reported cognitive function, and depression. Background characteristics and relevant clinical history will be obtained through an enrollment survey and chart review. The primary aim of the study is to describe the prevalence and extent of cognitive impairment in ITP and explore associated risk factors. This study will also assess the feasibility of longitudinal cognitive testing in patients with ITP and describe any observed changes in cognition over time.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years
* A clinical diagnosis of persistent or chronic ITP, as defined by a history of platelet counts <50 x 109/L on two occasions in the preceding 3 to 12 months or >12 months, respectively, and documented response to at least 1 prior ITP-directed therapy. ITP-directed therapies include corticosteroids, intravenous immune globulin, Rho(D) immune globulin, splenectomy, thrombopoietin receptor agonists, and fostamatinib. Other qualifying agents used for the treatment of ITP are permissible with approval of the principal investigator.
* Ability to follow instructions in English.

Exclusion Criteria:

* Pre-existing diagnosis of cognitive impairment from dementia, stroke, or other neurologic disease.
* Active psychiatric disorder, defined as uncontrolled major depression, schizophrenia, severe anxiety, or active alcohol or drug abuse.
* Active malignancy, requiring or likely to require chemotherapeutic or surgical treatment, except for non-melanoma skin cancer.
* Brain tumor or cranial surgery within the past year.
* Significant hearing or vision impairment that would preclude the ability to complete neurocognitive testing via a virtual platform.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a history of chronic or persistent ITP without pre-existing diagnosis of cognitive impairment will be recruited from the outpatient non-malignant hematology clinic at Massachusetts General Hospital (MGH).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Impairment of fluid cognition | Baseline
  Proportion of subjects with mild (T-score 1 to 2 standard deviations [SDs] below the normative mean) or major (>2 SDs below the normative mean) impairment of the composite measure of fluid cognition, as detected on the NIH Toolbox cognition battery.

SECONDARY OUTCOMES:
Feasibility of longitudinal assessments | 2 years
  Completion of annual study visit by at least 50% of the enrolled study population over course of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Mass General Brigham encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee.

REFERENCES:
- [Background] Frith J, Watson S, Bolton Maggs PH, Newton JL. Cognitive symptoms are common in immune thrombocytopenia and associate with autonomic symptom burden. Eur J Haematol. 2012 Mar;88(3):224-8. doi: 10.1111/j.1600-0609.2011.01730.x. Epub 2011 Dec 12. PMID 22044734
- [Background] Mitchell E, Frith J, Newton J. Fatigue and cognitive impairment in immune thrombocytopenic purpura remain stable over time: short report from a longitudinal study. Br J Haematol. 2019 Sep;186(5):777-781. doi: 10.1111/bjh.15993. Epub 2019 May 23. PMID 31119732
- [Background] Kuter DJ, Khan U, Maruff P, Daak A. Cognitive impairment among patients with chronic immune thrombocytopenia. Br J Haematol. 2024 Jul;205(1):291-299. doi: 10.1111/bjh.19495. Epub 2024 May 9. PMID 38724473